CLINICAL TRIAL: NCT01834391
Title: Diagnosis of Subclinical Urinary Tract Infections Using Advanced Microbiome Survey Techniques in High Risk Trauma Patients
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: J. Craig Venter Institute (Other)
Responsible Party: Principal Investigator, Martin D. Zielinski, Assistant Professor of Surgery, Mayo Clinic
Other Study IDs: 12-010185
Record Dates: First submitted 2013-03-20; First posted 2013-04-17 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Urinary Tract Infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Geriatric Traumatic Injury: Geriatric trauma pateints being admitted to Saint Marys Hosptial.

SUMMARY:
The purpose of this study is to see if the investigators can identify early those patients who are admitted to the hospital and have a urinary tract infection (UTI) or those patients that develop a UTI during their hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old or older admitted as a result of trauma to Saint Marys Hospital at Mayo Clinic

Exclusion Criteria:

* Prisoners
* Pregnancy
* Active urinary tract stones
* Less than 65 years of age

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Geriatric traumatic injury patients that were admitted to Saint Marys Hospital.
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Identify of bacteria, genes and proteins that are highly predictive of UTI development | Nine months
  To identify which bacteria, genes and proteins will be highly predictive of UTI development in geriatric trauma patients. We hypothesize that the combination of 16S rDNA and metaproteomics will identify the most informative biosignatures (species/genes/proteins) discerning UTI from asymptomatic bacteriuria.

SECONDARY OUTCOMES:
Biomarker candidates for UTIs recalcitrant to antibiotic treatment. | Nine months
Morbidity | 9 months
Mortality | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Zielinski, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States